CLINICAL TRIAL: NCT06214104
Title: Acupressure Therapy Method Applied in Newborn Heel Blood Collection and Fetus Effect of Position on Pain and Physiological Parameters
Brief Title: Acupressure Therapy Method and Heel Blood Effect of Position on Pain and Physiological Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: ETK00-2023-0237; Hulya Fırat Kılıc (Other: Eastern Mediterranean University)
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Newborn; Vitality
Keywords: Newborn, heels lancet, acupressure, fetal position

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- acupressure (Experimental): Acupressure Massage; It will be applied to BL 60 and K3 areas. The application will be applied in successive pressures with the thumb on each point for an average of 45-60 seconds.
  Interventions: Behavioral: Acupressur
- fetal position (Experimental): The fetal position will be given with the newborn in the right side position, with the arms and legs joined in the midline.
  Interventions: Behavioral: Acupressur
- Control group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Acupressur — Acupressure Massage; It will be applied to BL 60 and K3 areas. The application will be applied in successive pressures with the thumb on each point for an average of 45-60 seconds.The fetal position will be given with the newborn in the right side position, with the arms and legs joined in the midline.
  Other Names: fetal position
  Arms: acupressure; fetal position

SUMMARY:
It is important that integrated methods, which will not have a negative impact on the future health of babies who have just started life, are used in neonatal pain management by nurses who are in direct contact with babies, in terms of their ease of applicability. In addition, considering that by reducing the pain of newborns, their comfort will increase, mother-baby bonding will be greater, the newborn's adaptation to the outside world will increase, and sensory neural development will be positively affected. It is important for shaping. When the literature was examined, no study was found that examined the effect of the acupressure therapy method applied during heel blood collection of newborns and the effect of the fetal position on pain together. Accordingly, our study aimed to investigate the effects of these two important methods on pain and physiological parameters in newborns.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), the neonatal period covers the first 28 days of life from birth. A healthy newborn; It is a baby born between 38-40 weeks of gestation in the uterus, who cries after birth, adapts easily to the outside world, and does not have physiological, pathological or neurological problems (Deniz, 2023). It is important to detect some diseases that can be diagnosed early in the neonatal period so that the baby can have a healthy later life (Perry, 2018). These diseases; phenylketonuria (PKU), congenital hypothyroidism (CH), biotinidase deficiency (BE), cystic fibrosis (CF), Congenital Adrenal Hyperplasia, and Spinal Muscular Atrophy (SMA) (TC Ministry of Health). When these diseases are diagnosed early, the damage that may occur in the newborn can be reduced or eliminated with the necessary treatment and precautions (İçke, 2017). Screenings are carried out as a public health measure all over the world and in our country to detect these diseases for early diagnosis in the neonatal period (TC Ministry of Health). Most of these diseases, determined by heel blood collection and laboratory examinations, can be detected within the first two weeks (Bayrak, and Ünsal, 2021). The best time to take a blood sample is between the 36th and 72nd hours after birth. In addition, it is preferred that the baby has been feeding for 48 hours in order to perform scans (Ovalı, 2019; Bayrak and Ünsal, 2022). Taking a heel blood sample is a painful procedure for newborns. In the past, it was accepted that newborns did not feel pain and did not remember pain experiences because they were biologically immature. However, in recent years, studies in this field have been carried out in the 20-24 weeks of fetal life. It has been shown that the patient has the ability to respond to pain starting from weeks (Inmakulada et al, 2023). Pain perception is affected by the age, developmental level, cognitive and communication skills of babies and children, as well as previous pain experiences and beliefs (Varela, 2014;). It is also reported that painful stimuli change the perception of pain in the long term, increasing chronic pain syndromes and somatic complaints, and causing learning disorders, behavioral problems and attention deficit in the future as a result of recurrent pain (Akcan.2017; Eroğlu, 2018; Kahraman,2020; Glenzel,2023). . In line with this information, importance has begun to be given to the pain management of newborn babies in the literature and scales that detect pain have been developed (Bucsea 2019; Karakoç and Aydın 2022; Glenzel, 2023; It is noteworthy that there are more pharmacological methods to reduce pain in newborns. However, pharmacological applications in newborns have side effects and newborns It has been shown in literature studies that it will have a negative effect on the patient (Akcan, Polat, 2017). For this reason, integrative treatment methods, which are widely used today, are more recommended for neonatal pain management (Guney, 2017). Because these methods are non-invasive and do not cause any side effects. Its use is more encouraged. When the literature is examined, the integrative methods used in heel blood collection include breastfeeding, fetal position, swaddling, pacifier giving, oral glucose, acupressure, foot reflexology, kangaroo care, breast milk smell, mother and father's voice, mother's heart sound, music, white noise, There are many methods such as amniotic fluid smell, lavender smell (Aygül.2023; Memiş, 2023; Atal, 2019; Kale, 2019; Şafak, 2021; Tuncay, 2020; Deniz, 2019; Oğul, 2018; Avçin, 2017). There have been studies reporting that these methods have various effects on pain in newborns (Glenzel, 2023; Karakoç, 2022; Ceylan, 2017).

It has been reported that acupressure application reduces pain and anxiety in newborns, especially due to invasive interventional procedures (Deniz, 2019). Acupressure reveals the body's self-healing mechanism by making biochemical changes in the body. Acupressure affects the pain mechanism by applying pressure to acupuncture points (Özkan and Balcı, 2018). When studies in the literature are examined, it is reported that acupressure applied during heel blood collection reduces the newborn pain score (Deniz, 2019). Another nonpharmacological method used to reduce pain is the fetal position. Fetal position; It is a sub-form of the method of taking the baby into the nest and is the process of keeping the baby's upper and lower extremities in flexion with the hand and placing the body in a closed position close to the midline. It is reported that this method activates the regulatory systems of babies by providing heat and tactile stimulation, blocks painful stimuli from the external environment and reduces the pain felt by the baby (Avçin, 2015; Kemer and İşler, 2020). In a study, the effect of the fetal position during heel blood collection on pain, heart rate and oxygen saturation was examined and it was reported that the average pain score of babies in the fetal position was lower (Kale, 2018). It is important that integrated methods, which will not have a negative impact on the future health of babies who have just started life, are used in neonatal pain management by nurses who are in direct contact with babies, in terms of their ease of applicability. In addition, considering that by reducing the pain of newborns, their comfort will increase, mother-baby bonding will be greater, the newborn's adaptation to the outside world will increase, and sensory neural development will be positively affected. It is important for shaping. When the literature was examined, no study was found that examined the effect of the acupressure therapy method applied during heel blood collection of newborns and the effect of the fetal position on pain together. Accordingly, our study aimed to investigate the effects of these two important methods on pain and physiological parameters in newborns.

ELIGIBILITY:
Inclusion Criteria:

* Birth week 38-40,
* Within the first fifteen days of postnatal
* Birth weight is 2500-4000 grams,
* whose general condition is stable,
* He is with his mother and is literate,
* Mothers and newborns who agreed to participate in the research.

Exclusion Criteria:

* In need of oxygen support,
* Fed by orogastric tube,
* In need of parenteral nutrition,
* Receiving analgesic treatment,
* Having physical, metabolic and genetic diseases,
* Before the procedure, the Neonatal Infant Pain Scale (NIPS) score is ≥ 3 and above,
* Newborns who were hospitalized in the neonatal intensive care unit

Ages: 1 Week to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale:NIPS | 5 month
  It is a scale whose validity and reliability was established by Lawrence in 1993 for preterm and term babies and is used to evaluate the pain experienced by the newborn until the 6th week. It was developed to evaluate the behavioral pain responses of newborn babies 2 minutes before invasive procedures, 5 minutes during the procedure, and 3 minutes after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Abic, 1, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF, CSR

REFERENCES:
- [Result] Lemus-Varela Mde L, Sola A, Golombek S, Baquero H, Borbonet D, Davila-Aliaga C, Del Moral T, Lara-Flores G, Lima-Rogel MV, Neira-Safi F, Natta D, Oviedo-Barrantes A, Rodriguez S; Consenso Clinico de Dolor y Estres Neonatal, de la Sociedad Iberoamericana de Neonatologia (SIBEN). [Consensus on the diagnostic and therapeutic approach to pain and stress in the newborn]. Rev Panam Salud Publica. 2014 Nov;36(5):348-54. Spanish. PMID 25604106
- [Result] Yilmaz D, Inal S. Effects of three different methods used during heel lance procedures on pain level in term neonates. Jpn J Nurs Sci. 2020 Oct;17(4):e12338. doi: 10.1111/jjns.12338. Epub 2020 Apr 2. PMID 32239753